CLINICAL TRIAL: NCT03518983
Title: Low-intensity Shockwaves Therapy: Validation of an Evidence Based Protocol in a Randomized, Sham-controlled Trial for the Treatment of Patients With Moderate Vasculogenic Erectile Dysfunction
Brief Title: Low-intensity Shockwaves Therapy for the Treatment of Patients With Moderate Vasculogenic Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, President, Institute for the Study of Urological Diseases Thessaloniki, Greece, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5142/2-4-18
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Group (Sham Comparator): The subjects of this group will receive shockwave treatments (12 sessions for all subjects, 5000 shockwaves at each session), twice a week (total of 6 weeks) by the sham probe.
  Interventions: Device: Dornier Aries2 device (sham probe)
- Active Group (Active Comparator): The subjects of this group will receive shockwave treatments (12 sessions for all subjects, 5000 shockwaves at each session), twice a week (total of 6 weeks) at energy level 7.
  Interventions: Device: Dornier Aries2 device

INTERVENTIONS:
Device: Dornier Aries2 device — The Dornier Aries2 device and will be used for the purpose of the study. LI-ESWT will be applied to the penile shaft and the 2 crura(two sites).
  Arms: Active Group
Device: Dornier Aries2 device (sham probe) — The Dornier Aries2 device and will be used for the purpose of the study but the active probe will be replaced by an identical sham probe.
  Arms: Sham Group

SUMMARY:
This is a double-blind, sham-controlled randomized, 2 parallel arms, clinical trial with a 12-month recruitment period. All patients will be PDE5I users/responders. After 1 month wash-out period, ED patients will be screened, in order to randomize 70 men with vasculogenic ED.Patients will be randomized in 2 groups (35 subjects in each group) to receive shockwave treatments (12 sessions for all subjects, 5000 shockwaves at each session), twice a week (total of 6 weeks) either at energy level 7 or at sham-control , without treatment interval. The IIEF-ED domain will be evaluated at Visit 1 and, consequently, at baseline and all follow up visits together with the SEP diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate.
2. Age 40-70 years.
3. Sexually active in a stable, heterosexual relationship of more than three months duration.
4. Presence of Erectile Dysfunction for at least 6 months.
5. At Screening, diagnosed as Vasculogenic erectile dysfunction based on sexual history
6. PDE5i users and report some or good response to PDE5i. Last reported PDE5i use must be within 30 days of Screening Visit.
7. Agree to suspend all ED therapy for the duration of the study.
8. Agree to attempt sexual intercourse at least 4 times during the last 4 weeks prior to Visit 2/Randomization, 1-month Follow Up and 3-month Follow-Up without being under the influence of alcohol or recreational drugs. Agree to document the outcome using the Sexual Encounter Profile (SEP) diary.
9. At Visit 2 (after PDE5i washout), SEP Q2, "Were you able to insert your penis into your partner's vagina?" answered "YES" 25% - 100% of the time.
10. At Visit 2, SEP Q3, "Did your erection last long enough for you to have successful intercourse?" answered "YES" 0% - 50% of the time.
11. At Visit 2, IIEF-EF score 11 - 16.

13. At Visit 2, IIEF Q3 score 2 - 5. 14. At Visit 2, IIEF Q4 score 1 - 3.

Exclusion Criteria:

1. Previous major pelvic surgery or pelvic trauma that could impact erectile function, such as radical prostatectomy, radical cystectomy, rectal surgery. Patients with previous TURP surgery without sequelae of iatrogenic ED, may be included.
2. Previous penile surgery of any kind except circumcision and condyloma removal, such as penile lengthening, penile cancer surgery, penile plication, grafting.
3. Previous history of priapism or penile fracture
4. Previous radiation therapy to pelvis.
5. Abnormal serum testosterone level defined as a value lower than 300 ng/dL (indicative of untreated hypogonadism), or greater than 1197 ng/dL.
6. Current or previous hormone usage, other than prescribed testosterone, clomiphene or thyroid medication. Subjects with prior or current use of hormonal treatment for prostate cancer are also excluded.
7. ED due primarily to psychogenic factors
8. Peyronie's Disease or penile curvature that negatively influences sexual activity.
9. Patients with cardiac or non-cardiac electrical devices implanted.
10. Open wound or any anatomical or neurological abnormalities in the treatment area.
11. Uncontrolled diabetes mellitus with glucose >200 mg/dL (once or more times/week during the last month prior to recruitment, or during screening blood test).
12. Patients with generalized polyneuropathy, or neurological conditions irrespective of cause, such as severe diabetes, multiple sclerosis or Parkinson's Disease.
13. Refusal to suspend ED therapy for duration of study. Subjects who are using Tadalafil as a treatment for BPH (Benign Prostatic Hyperplasia) will also be excluded.
14. Men deemed not healthy enough to participate in sexual activity.
15. Any condition or behavior that indicates to the Principal Investigator that the subject is unlikely to be compliant with study procedures and visits.
16. Any health history or laboratory result that indicates to the Principal Investigator that the subject has a significant medical condition and should not participate in the study.
17. Known allergy to ultrasound gel.
18. History of consistent treatment failure with PDE5 inhibitors for therapy of ED.
19. Any history of significant psychiatric disease, such as bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity. Patients who are currently using SSRI or psychotropic medications e.g., Citalopram (Celexa), Escitalopram (Lexapro, Cipralex), Paroxetine (Paxil, Seroxat), Fluoxetine (Prozac), Fluvoxamine (Luvox, Faverin),Sertraline (Zoloft, Lustral), Clonazepam (Klonopin), Alprazolam (Xanax), Aripiprazole (Ambilify), Clozapine (Clozaril), Risperidone (Risperdal), Quetiapine (Seroquel), Olanzapine (Zyprexa) are also excluded.
20. Partners who are < 18 years of age, who are nursing, who are known to be pregnant at screening, who wish to become pregnant during the study period, who have any gynecologic problems, sexual dysfunction, or major medical conditions that would limit participation in sexual intercourse.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
The difference between the 2 groups in the percent of subjects who achieve clinically important difference (MCID) in the EF domain score of the IIEF | at 3 month follow up visit
  MCID is defined according to baseline ED severity as:Improvement by 5 or more in the EF domain score of the IIEF for patients with moderate ED(EF scores 11-16) at baseline

SECONDARY OUTCOMES:
The difference between the 2 groups in the change of the EF domain score of the IIEF | baseline and 3 month follow up visit.
  EF domain of the IIEF questionnaire will be completed
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline and 3 month follow up visit.
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported
Number of patients with treatment related adverse events | 18 weeks
  Potential treatment related adverse events after the first LI-ESWT session and during the 3 month follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Hatzichristou, Prof., Principal Investigator — G.Gennimatas General Hospital, Thessaloniki,Greece
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalyvianakis D, Memmos E, Mykoniatis I, Kapoteli P, Memmos D, Hatzichristou D. Low-Intensity Shockwave Therapy for Erectile Dysfunction: A Randomized Clinical Trial Comparing 2 Treatment Protocols and the Impact of Repeating Treatment. J Sex Med. 2018 Mar;15(3):334-345. doi: 10.1016/j.jsxm.2018.01.003. Epub 2018 Feb 1. PMID 29396020
- [Background] Kalyvianakis D, Hatzichristou D. Low-Intensity Shockwave Therapy Improves Hemodynamic Parameters in Patients With Vasculogenic Erectile Dysfunction: A Triplex Ultrasonography-Based Sham-Controlled Trial. J Sex Med. 2017 Jul;14(7):891-897. doi: 10.1016/j.jsxm.2017.05.012. PMID 28673433